CLINICAL TRIAL: NCT00661544
Title: Phase I/II Study of the Combination of Arsenic Trioxide With Ascorbic Acid and High-Dose Melphalan for Patients With Multiple Myeloma
Brief Title: Arsenic Trioxide With Ascorbic Acid and Melphalan for Myeloma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0603
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Results first posted 2009-07-14 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Multiple Myeloma; Stem Cell Transplantation
Keywords: Multiple Myeloma; Ascorbic Acid; Vitamin C; Arsenic Trioxide; Trisenox; Melphalan; Autologous Stem Cell Transplant; Stem Cell Transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Arsenic Trioxide; Melphalan; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arsenic Trioxide + Vitamin C + Melphalan (Experimental): Arsenic Trioxide + Ascorbic Acid + Melphalan as a preparative regimen for autologous stem cell transplantation (delivered on Day 0)
  Interventions: Drug: Arsenic Trioxide; Drug: Melphalan; Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Arsenic Trioxide — Dose Level 1: None; Dose Level 2: 0.15 mg/kg days Intravenous (IV) Days -9 to -3; Dose Level 3: 0.25 mg/kg days IV Days -9 to -3.
  Other Names: Trisenox
Drug: Melphalan — Dose Levels 1, 2, & 3: 100 mg/m2 IV Days -4, -3.
Drug: Ascorbic Acid — Dose Levels 1, 2, & 3: 1000 mg IV Days -9 to -3.
  Other Names: Vitamin C

SUMMARY:
1. To evaluate the toxicity and safety of a combination of arsenic trioxide with ascorbic acid and high-dose Melphalan in patients with multiple myeloma
2. To evaluate the efficacy of a combination of arsenic trioxide with ascorbic acid and high-dose Melphalan in patients with multiple myeloma
3. To determine the effects of arsenic trioxide on melphalan pharmacokinetics

DETAILED DESCRIPTION:
Treatment:

High-dose melphalan followed by a transplant of autologous stem cells is thought to be one of the most effective ways to treat multiple myeloma. However, the number one cause of treatment failure in these patients is the disease coming back.

High-dose melphalan has been used in multiple myeloma for more than two decades and is considered the standard of care for this disease. Recent research in the laboratory and clinical trials has shown that Arsenic trioxide is an effective treatment against multiple myeloma. It leads to tumor cell death in myeloma cell lines and in myeloma patients. Arsenic trioxide can also make melphalan a more effective antimyeloma agent. This research has also shown that vitamin C enhances the anti-myeloma activity of arsenic trioxide by making it more toxic to myeloma cells. The purpose of this study is to learn if a combination of arsenic trioxide, vitamin C, and melphalan will be safe, well-tolerated and effective in myeloma patients.

Before treatment begins, you will have several tests performed to study the status of the disease before you begin taking the study medication. You will have a bone marrow aspirate and biopsies. An aspirate is the drawing of liquid marrow with a syringe, while a biopsy is the removal of a small core of bone with a hollow needle. Aspirate can be done from the hip bone or chest, while biopsy is always from the hip bone. You will have cytogenic tests, to see if there are any genetic abnormalities in your DNA. You will have a bone survey done, where the doctor will look at X-rays of your bones for any myeloma-related bone changes.

You will have routine and specialized blood tests done (about 2 tablespoons), to measure blood counts, platelets, blood clotting, kidney function, electrolyte counts, and levels of disease in your blood. You will also have a urine test to measure level of myeloma in your urine. You will have a pulmonary function test, to check if your lungs is strong enough to withstand high-dose chemotherapy. You will have an initial electrocardiogram (EKG) and also a MUGA scan that will measure how strong your heart functions are.

Women who are able to have children must have a negative blood pregnancy test before participating in this study.

If you agree and are eligible, you will be assigned to receive one of 3 arms. In the first arm only melphalan and vitamin C, but no Arsenic trioxide will be given. In the second and third arms, doses of arsenic trioxide together with Vitamin C and melphalan will be given. Not all patients in this study will get the same dose of arsenic. Your dose assignment will depend on the experience of other patients with this combination. The first 3 patients on this study will get the lowest dose of arsenic trioxide.

Arsenic trioxide will be given through a needle in the vein over a period of 2 hours, once a day for 7 days. At the same time, vitamin C will be given once a day through the vein for 7 days. On the last 2 days of arsenic trioxide treatment, melphalan will be given through the vein over one hour after the arsenic. You will have your stem cells reinfused 2 days after the last dose of melphalan.

Some patients agreeing to the optional procedure will receive one of the doses of melphalan before starting the arsenic.

You will receive standard inpatient and outpatient transplant care and testing. This involves blood and bone marrow tests, heart tests, lung tests and x-rays before the study drug treatment and the transplant. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Blood tests (about two tablespoons) will be drawn at least once a week for the first month after the transplant, and then once every month for the next 3 months.

Bone marrow biopsies and tests to check the level of myeloma protein in the urine and the blood are also performed at 3, 6 and 12 months after the transplant.

You will be taken off study one year after transplant, if your disease does not come back. Patients off study will still return for their routine post-transplant follow up visits as decided by their transplant physician. If your disease comes back or intolerable side effects occur, you will be taken off study.

This is an investigational study. Both arsenic trioxide and melphalan are commercially available and have been approved for use in patients with myeloma, though their use together with vitamin C is investigational. About 32 patients are expected to participate in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Multiple Myeloma in any of the following disease categories: a) Primary Refractory Disease b) Consolidation of a partial remission (defined as a decrease but continued presence of monoclonal protein on serum and urine immunofixation electrophoresis, and/or the presence of plasmacytosis on bone marrow aspirate and biopsy) c) All patients relapsing after prior therapy .
2. Age up to 70 years.
3. Zubrod Performance Status (PS) of <2.
4. Left ventricular ejection fraction >40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
5. Forced vital capacity (FVC); Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and Carbon Monoxide Diffusing Capacity (DL CO) >40%. No symptomatic pulmonary disease.
6. Serum bilirubin <2 times upper limit of normal, SGPT <4 times upper limit of normal. No evidence of chronic active hepatitis or cirrhosis. No effusion or ascites >1L prior to drainage.
7. HIV-negative.
8. Patient is not pregnant.
9. Patient or guardian able to sign informed consent.
10. Corrected QT interval less than 500 msec.

Exclusion Criteria:

1. Corrected QT interval greater than 500 msec
2. Patients in complete remission (defined as the absence of monoclonal protein on serum and urine immunofixation electrophoresis, and the absence of plasmacytosis in bone marrow aspirate and biopsy).
3. Patients with non-secretory myeloma.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar H. Qazilbash, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 03/31/2004 through 08/02/2005. All pariticipants recruited at U.T. M.D. Anderson Cancer Center.
Period: Overall Study
Arm/Group | Arsenic Trioxide + Vitamin C + Melphalan
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arsenic Trioxide + Vitamin C + Melphalan
Number analyzed (Participants) | 48
Age, Customized [Median (Full Range); unit: years] | 54 [35 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Bone marrow aspirate and biopsy performed to assess complete response and overall response rate.
Time Frame: 3, 6 and 12 months
Measure: Number; unit: Participants
Arm/Group | Arsenic Trioxide + Vitamin C + Melphalan
Number analyzed (Participants) | 48
Participants
  Complete Response | 11
  Overall Response (Complete + Partial Response) | 36

ADVERSE EVENTS:
Time Frame: 3 years and 1 month
Arm/Group | Arsenic Trioxide + Vitamin C + Melphalan
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No